CLINICAL TRIAL: NCT00028015
Title: A Phase II Study of Second-Line SarCNU (NSC 364432) in Patients With Recurrent/Metastatic Colorectal Cancer
Brief Title: SarCNU in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I146; CAN-NCIC-IND146 (Other: PDQ); CDR0000069113 (Other: PDQ)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — 2-((((2-chloroethyl)nitrosoamino)carbonyl)amino)propanamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: SarCNU

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of sarCNU in treating patients who have recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of SarCNU in patients with recurrent or metastatic colorectal cancer.
* Determine the qualitative and quantitative toxicity of this drug in these patients.
* Determine the time to progression and survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral SarCNU on days 1, 5, and 9. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response (CR) receive 2 additional courses beyond documentation of CR. Patients who achieve partial response (PR) receive 4 additional courses beyond documentation of PR.

Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 6-8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Locally recurrent or metastatic disease
  * Previously treated with 1 chemotherapy regimen for recurrent or metastatic disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * No prior radiotherapy to indicator lesion (clear disease progression or new lesion within a prior radiation port is acceptable)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 120,000/mm^3

Hepatic:

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary:

* DLCO at least 80% predicted
* FVC at least 80% predicted
* No history of significant pulmonary disease
* No concurrent symptomatic pulmonary disease (e.g., chronic obstructive pulmonary disorder, chronic asthma)

Other:

* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No other serious illness or medical condition that would preclude study
* No ongoing or active uncontrolled infection
* No history of significant neurologic or psychiatric disorder that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* Prior adjuvant chemotherapy allowed
* No prior nitrosoureas
* No prior second-line chemotherapy for recurrent or metastatic disease
* At least 4 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy as part of primary therapy allowed
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Prior surgery as part of primary therapy allowed
* Prior reoperation for recurrent disease allowed
* At least 2 weeks since prior surgery other than biopsy

Other:

* At least 4 weeks since prior investigational agent
* No other concurrent investigational agents or therapy
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2001-10-30 (Actual); Primary Completion 2003-09-22 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph PW Wong, MD, FRCPC, Study Chair — CancerCare Manitoba
Locations (7):
- Canada (7):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre- Dame du CHUM, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wong RP, Baetz T, Krahn MJ, Biagi J, Wainman N, Eisenhauer E; National Cancer Institute of Canada Clinical Trials Group. SarCNU in recurrent or metastatic colorectal cancer: a phase II study of the National Cancer Institute of Canada Clinical Trials Group. Invest New Drugs. 2006 Jul;24(4):347-51. doi: 10.1007/s10637-006-5730-2. PMID 16502354